CLINICAL TRIAL: NCT04014842
Title: Post-Approval Study for Reconfirmation Analysis Mode Algorithm
Brief Title: RapidShock Post-Approval Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12701
Record Dates: First submitted 2019-04-25; First posted 2019-07-10 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- RapidShock (Other): Patients receiving xseries device with rapid shock enabled
  Interventions: Device: RapidShock

INTERVENTIONS:
Device: RapidShock — Use of the Reconfirmation Analysis Mode algorithm

SUMMARY:
Compare the performance of the Reconfirmation Analysis Mode algorithm to the performance goals recommended by the American Heart Association.

ELIGIBILITY:
Inclusion Criteria:

* 8 years of age or older and weight ≥ 55 lbs (25 kgs)
* Out-of-hospital cardiac arrest (OOHCA)
* Non-traumatic cardiac arrest

Exclusion Criteria:

* Weight less than 55 lbs (25 kgs)
* Do not attempt resuscitation (DNAR) orders

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2756 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Algorithm accuracy | average of up to 1 hour after device placement
  Accuracy of the algorithm compared to manual annotation for each rhythm

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Ventura County Fire Department, Camarillo, California
  - Colorado Springs Fire Department, Colorado Springs, Colorado
  - East Baton Rouge Parish EMS, Baton Rouge, Louisiana
  - Detroit Fire Department, Detroit, Michigan
  - M Health Fairview EMS, Saint Paul, Minnesota
  - Fort Worth Fire Department, Fort Worth, Texas
  - San Antonio Fire, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No